CLINICAL TRIAL: NCT00140283
Title: Phase IV Cluster Randomised Controlled Trial With 2 Parallel Groups, to Evaluate the Effectiveness of a Educational Intervention to Improve the Resolution Capacity.
Brief Title: Effectiveness of a Educational Intervention to Improve the Resolution Capacity of Primary Health Care Teams.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Catalan Institute of Health (Other Government)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: PI031409; P03/30
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2005-09-01 (Estimated); Status verified 2005-08

CONDITIONS: Referral and Consultation
Keywords: Effectiveness; Educational intervention; Primary health care

INTERVENTIONS:
Procedure: Educational interactive intervention

SUMMARY:
There is a great variability in the different primary care teams referral rate. And variability means inappropriateness somewhere in the process of care. The most important determinants of the variability are the attitude and knowledge of the professional, the existence and availability of evidence, the resources available and the professionals practice style. To improve the knowledge of the professionals could be a way to decrease the variability. Because of this, we have the aim to determinate the effectiveness of an educational intervention to improve the primary care teams from the city of Barcelona referral rate.

DETAILED DESCRIPTION:
The aim of our study is to determinate if an active educational intervention (interactive sessions discussing clinical cases plus the minimal intervention) reduces the professionals referral rate compared with the minimal intervention group (written adapted clinical practice guidelines and feedback about their referral rate compared with other primary care teams). It is a cluster-randomized controlled trial stratified by the percentage of reform and the referral rate. The subjects were primary care physicians of the 51 teams of Barcelona city attending 1.160.748 inhabitants.

ELIGIBILITY:
Inclusion Criteria:

* Primary care teams who agree to participate.
* Primary care teams attending adult population (older than 14).

Exclusion Criteria:

* Primary care teams where the intervention would be difficult to take place.
* Primary care teams where the referral rate is not available.
* Primary care teams with a percentage of reform lower than 40%.

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 48
Dates: Start 2004-07; Study Completion 2005-05

PRIMARY OUTCOMES:
Total number of referrals of the selected condition done by the primary care professionals to specialized consultants by 100 patients attended in 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Casajuana, Physician, Principal Investigator — Catalan Institute of Health
Locations (1):
- Àmbit Barcelona (Catalan Institute of Health), Barcelona, Barcelona, Spain